CLINICAL TRIAL: NCT04040530
Title: Patient Reported Outcome After Nephron Sparing Treatment of Small Renal Tumours
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Region of Southern Denmark (Other)
Collaborators: University of Southern Denmark (Other); Region Zealand (Other)
Responsible Party: Principal Investigator, Theresa Junker, Principal Investigator, Region of Southern Denmark
Other Study IDs: Nephspare PRO
Record Dates: First submitted 2019-06-25; First posted 2019-07-31 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Renal Cell Carcinoma; Quality of Life
Keywords: Renal Cell Carcinoma; Nephron sparing treatment; Quality of life; Patient Reported Outcome Measures; Kidney Neoplasms; Cryosurgery
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cryoablation: Consecutive patients diagnosed with biopsy proven renal cell carcinoma at stadium T1a or T1b, from the Region of Southern Denmark or Region Zealand, treated with CT-guided cryoablation at Odense University Hospital in the period from 1/6-2019 to 1/6-2021.
  Interventions: Procedure: CT-guided cryoablation
- Partial nephrectomy: Consecutive patients diagnosed with biopsy proven renal cell carcinoma at stadium T1a or T1b, from the Region of Southern Denmark or Region Zealand, treated with partial nephrectomy at Odense University Hospital or Zealand University Hospital in the period from 1/6-2019 to 1/6-2021.
  Interventions: Procedure: Partial nephrectomy

INTERVENTIONS:
Procedure: CT-guided cryoablation — Percutaneous computed tomography guided cryoablation with the patient in sedation or general anaesthesia.
  Groups: Cryoablation
Procedure: Partial nephrectomy — Surgical removal of the renal cancer, leaving the healthy renal tissue. Surgery is either done laparoscopically, robot-assisted laparoscopically or as an open surgery. The patient is under general anaesthesia.
  Groups: Partial nephrectomy

SUMMARY:
The present study is an observational study designed to assess and compare clinical outcome and quality of life after nephron sparing treatment of small renal tumors.

Partial nephrectomy, where the tumor is being be surgically removed, has traditionally been the preferred nephron sparing treatment for small renal cell carcinomas (RCC). Cryoablation was introduced 20 years ago as a treatment option for patients with RCC with a high surgical risk. Previously, this group of patients had no available treatment. Cryoablation is a minimally invasive treatment that uses extreme cold to destroy the cancer. In recent years, indications for cryoablation of RCC has extended. Cryoablation is now offered as a curative treatment, also including patients without severe comorbidity.

Retrospective studies imply that patients with RCC have lower quality of life compared to other cancers and that choice of treatment and remaining healthy renal tissue have a correlation with quality of life. Knowledge about the patient perspective is crucial in relation to delivering the highest quality of care in the healthcare system. Exploring quality of life through patient reported outcome is one way of exploring the patient perspective.

In this prospective study the investigators aim to assess clinical outcome and quality of life after partial nephrectomy and cryoablation. Results are expected to generate evidence-based knowledge essential in treatment decisions for RCC globally.

DETAILED DESCRIPTION:
The overall aim of this prospective study is to assess and compare clinical outcome and health related quality of life after partial nephrectomy and cryoablation of renal tumors at stadium T1 in adult patients. The specific objectives is:

* To describe treatment characteristics (treatment type, knife time, type of anaesthesia) with i) cryoablation and ii) partial nephrectomy on patients with T1 renal tumors in the Regions of Southern Denmark and Zealand.
* To describe self-reported health related quality of life in adult patients with T1 renal tumors undergoing i) cryoablation and ii) partial nephrectomy in the Regions of Southern Denmark and Zealand.
* To compare patient and tumor characteristics (age, sex, BMI, performance status, American Society of Anaesthesiologists' (ASA) classification group, comorbidity, other cancer diagnosis, smoking and alcohol use, tumor location and size, and tumor histology) in patients with T1 renal tumors treated with i) Cryoablation or ii) partial nephrectomy in the Regions of Southern Denmark and Zealand.
* To compare complications, length of hospital stay, treatment success within follow-up, readmission rate and in-hospital mortality after after i) cryoablation and ii) partial nephrectomy of renal tumors at stadium T1 in adult patients in the Regions of Southern Denmark and Zealand.
* To compare self reported quality of life after i) cryoablation and ii) partial nephrectomy of renal tumors at stadium T1 in adult patients in the Regions of Southern Denmark and Zealand.
* To identify potential patient or tumor characteristics reducing quality of life after i) cryoablation and ii) partial nephrectomy of renal tumors at stadium T1 in adult patients in the Regions of Southern Denmark and Zealand.

All eligible patients will be offered inclusion. Patients will be allocated to treatment group based on shared decision making between the patient and the treating urologist and recommendation from a multidisciplinary team conference. This reflecting the clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing CT-guided cryoablation of histologically verified primary renal cancer at stage T1
* Patients undergoing partial nephrectomy of histologically verified primary renal cancer at stage T1
* Patients who understand and read Danish.

Exclusion Criteria:

* Patients diagnosed with dementia.
* Patients with tumours > 7 cm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are recruited from the Department of Urology at Odense University Hospital and Zealand University Hospital based in The Region of Southern Denmark and Region Zealand respectively. Odense University Hospital and Zealand University Hospital are the only centers offering nephron sparing treatment for renal cell carcinomas within the two regions.
  The Region of Southern Denmark and Region Zealand are two out of the five regions in Denmark. They have a population of about 2 million people combined. The population of the regions are considered demographic comparable.
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2019-06-07 (Actual); Primary Completion 2021-02-07 (Actual); Study Completion 2026-02-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in health-related Quality of life measured by the validated Danish version of The European Organisation for Research and Treatment of Cancer - Core Quality of Life Questionnaire (EORTC QLQ C-30) | Change from baseline at 14 days and 3 months postoperatively.
  EORTC QLQ C- 30 will be used for quality of life measurement. A scale range 0-100, a higher score indicating better quality of life within five functional scales ( physical, role, cognitive, emotional, and social), three symptom scales (fatigue, pain, and nausea and vomiting), a global health status scale and the following six single item symptom measures; dyspnea, insomnia, appetite loss, constipation, diarrhea, and functional difficulties.
Change from baseline in health-related Quality of life (HRQoL) to 3 months after treatment measured by the validated Danish version of SF-12v2. | 3 months
  HRQoL will be assessed by the Short Form 12 version 2.0 (SF-12v2) Health Survey scores.
Self evaluation of rehabilitation and experience of course of treatment measured by a locally validated questionnaire. | 3 months
  Patients' self evaluation of rehabilitation and course of treatment will be assessed by the locally validated rehabilitation questionnaire for renal cancer (RQRC). The questionnaire consists of seven items. Responses will be reported in percentages.
Number of participants with treatment related complications within the first 30 days after treatment. | 30 days
  Graded and classified according to the Clavien-Dindo classification.
Number of participants with treatment related complications between 30 and 90 days after treatment. | From 30 to 90 days postoperatively
  Graded and classified according to the Clavien-Dindo classification.
Number of participants who are readmitted to the hospital after discharge from treatment. | Within the first 30 days postoperatively
  Readmission to the hospital after discharge
Treatment success | 3 months
  The degree of incomplete ablation after cryoablation, visualized on CT, in comparison with the degree of positive surgical margin after partial nephrectomy, from histopathology.

SECONDARY OUTCOMES:
Length of hospital stay after nephron sparing treatment | up to 90 days
  Absolute number of days the patient is hospitalized after treatment.
Rate of in-hospital mortality | up to 90 days
  Mortality under hospitalization after initial treatment
Rate of cancer related mortality | Minimum of 3 months follow-up and up to 5 years.
  Cancer related mortality calculated from the date of treatment, to the date of death related to renal cell carcinoma or censored at the date at last follow-up.
Change from baseline in health-related Quality of life measured by the validated Danish version of EORTC QLQ C-30. | Change from baseline at 1-5 years postoperatively.
  The European Organisation for Research and Treatment of Cancer - Core Quality of Life Questionnaire (EORTC QLQ C-30) will be used for quality of life measurement. A scale range 0-100, a higher score indicating better quality of life within five functional scales ( physical, role, cognitive, emotional, and social), three symptom scales (fatigue, pain, and nausea and vomiting), a global health status scale and the following six single item symptom measures; dyspnea, insomnia, appetite loss, constipation, diarrhea, and functional difficulties.
Change from baseline in health-related Quality of life (HRQoL) measured by the validated Danish version of SF-12v2. | Change from baseline at 1-5 years postoperatively.
  HRQoL will be assessed by the Short Form 12 version 2.0 (SF-12v2) Health Survey scores.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Junker, PhD-student, Principal Investigator — Region of Sourthern Denmark, Odense University Hospital; Ole Graumann, MD, PhD, Study Director — Region of Sourthern Denmark, Odense University Hospital
Locations (2):
- Denmark (2):
  - Odense University Hospital, Odense C
  - Zealand University Hospital, Roskilde

IPD SHARING:
Plan to Share IPD: No